CLINICAL TRIAL: NCT01393808
Title: A Prospective, Randomized, Cross-over, Double-blind, Placebo-controlled Study to Assess the Antiproteinuric Effect of Selective Vitamin d Receptor Activation by Paricalcitol in Type 2 Diabetes Patients on Low or High Sodium Diet and Stable Ras Inhibitor Therapy
Brief Title: Salt Intake and Antiproteinuric Effect of Paricalcitol in Type 2 Diabetes
Acronym: PROCEED
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PROCEED; 2011-001713-14 (EudraCT Number)
Record Dates: First submitted 2011-07-12; First posted 2011-07-13 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes; Paricalcitol; Proteinuria; Sodium intake
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Proteinuria | interventions — paricalcitol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paricalcitol (Experimental)
  Interventions: Drug: Paricalcitol
- placebo (Placebo Comparator)
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Paricalcitol — 1-month Paricalcitol 2mcg/day
  Arms: Paricalcitol
Other: placebo — 1-month Placebo Treatment
  Arms: placebo

SUMMARY:
Proteinuria is an independent risk factor for cardiovascular morbidity and mortality and for renal disease progression. More proteinuria is associated with faster progression, whereas treatments that reduce proteinuria are renoprotective in both diabetic and non diabetic chronic kidney disease. Of note, lower the residual proteinuria achieved by treatment slower is the disease progression in the long term. On the basis of the above findings, proteinuria has become a target of renoprotective therapy.

Among different antihypertensive medications, those that inhibit the Renin Angiotensin System, such as angiotensin converting enzyme (ACE)inhibitors and angiotensin receptor blockers (ARBs), are those that at comparable blood pressure control, more effectively reduce proteinuria and slow renal disease progression. Thus they have become the key component of renoprotective therapy in patients with proteinuric chronic kidney disease. Observational studies found that their effectiveness, however, is limited or even fully blunted in patients who eat large amount of salt.

Experimental evidence indicates a renoprotective role of the vitamin D system in chronic renal disease. A recent randomized, controlled trial, add-on therapy with selective Vitamin D receptor activator paricalcitol showed an additive antiproteinuric effect in subjects with type 2 diabetes and chronic kidney disease on background Renin-angiotensin-system inhibitor therapy. This effect, however, was largely restricted to subjects with daily sodium intake exceeding 12 grams and was negligible in those with lower sodium intake. Thus, treatment with paricalcitol appears to be effective in particular in those patients who do not appreciably benefit of renin angiotensin system (RAS) inhibitors therapy because of high salt intake. Thus, whether the antiproteinuric effect of paricalcitol is modified by concomitant salt intake in patients with chronic kidney disease (CKD) on background RAS inhibitors therapy, is worth investigating.

The broad aim of this study is to evaluate the interaction between paricalcitol therapy and sodium intake in type 2 diabetes patients with proteinuric kidney disease on stable background RAS inhibitor therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients;
* Age > 18 years;
* Type 2 diabetes patients on low or high sodium diet and stable RAS inhibitor therapy with the following conditions:

Urinary albumin excretion (UAE) rate >300mg/24 hours (200 mcg/min); Serum creatinine <2 mg/dL, PTH ≥ 20 mEq/L and <110 mEq/L; Calcium and phosphorus levels < 9.5 mg/dl and < 5mg/dl, respectively; Controlled BP (systolic/diastolic <140/90 mmHg) while on stable RAS inhibitor therapy;

- Written informed consent.

Exclusion Criteria:

* Previous Vitamin D or Vitamin D analogs therapy (within 3 months prior to the study entry);
* Evidence of toxicity to Vitamin D;
* History of kidney stones;
* Poorly controlled Diabetes: Hb1Ac > 12%;
* Therapy with calcitonin, bisphosphonates, cinacalcet, glucocorticoids, immunosuppressive drugs or other drug that may affect calcium or bone metabolism;
* Cancer and any severe systemic disease or clinical condition that may jeopardize data interpretation or completion of the study;
* Any clinically relevant conditions that might affect study participation and/or study results;
* Any contraindication to be exposed to Paricalcitol;
* Pregnancy or lactating;
* Women of childbearing potential without following a scientifically accepted form of contraception;
* Legal incapacity.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2011-09; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Changes in urinary albumin excretion from baseline at 4 month. | At baseline and 1,2,3 and 4 month.

SECONDARY OUTCOMES:
Ambulatory and 24-hour blood pressure profile. | At 1 month.
Ambulatory and 24-hour blood pressure profile. | At 2 month.
Ambulatory and 24-hour blood pressure profile. | At 3 month.
Ambulatory and 24-hour blood pressure profile. | At 4 month.

CONTACTS AND LOCATIONS:
Locations (6):
- Italy (6):
  - Azienda Ospedaliera Ospedali Riuniti di Bergamo, Bergamo, Bergamo
  - ASL of Ponte San Pietro - Diabetologic Unit, Brembate, Bergamo
  - Clinical Research Center fo Rare Diseases Aldo and Cele Daccò, Ranica, Bergamo
  - Azienda Ospedaliera di Treviglio e Caravaggio - Unit of Diabetology and Metabolic Diseases, Romano di Lombardia, BG
  - Azienda Ospedaliera Bolognini - Unità di Medicina, Seriate, BG
  - Azienda Ospedaliera di Treviglio e Caravaggio - Unit of Diabetology and Metabolic Diseases, Treviglio, BG

REFERENCES:
- [Derived] Hodson EM, Cooper TE. Altered dietary salt intake for preventing diabetic kidney disease and its progression. Cochrane Database Syst Rev. 2023 Jan 16;1(1):CD006763. doi: 10.1002/14651858.CD006763.pub3. PMID 36645291
- [Derived] Prabhu RA, Saraf K. Vitamin D in diabetic nephropathy. J Postgrad Med. 2018 Jan-Mar;64(1):5-6. doi: 10.4103/jpgm.JPGM_311_17. No abstract available. PMID 29386411
- [Derived] Parvanova A, Trillini M, Podesta MA, Iliev IP, Ruggiero B, Abbate M, Perna A, Peraro F, Diadei O, Rubis N, Gaspari F, Carrara F, Stucchi N, Belviso A, Bossi AC, Trevisan R, Remuzzi G, de Borst M, Ruggenenti P; PROCEED Study Organization and the Scientific Writing Academy (SWA) 2016. Moderate salt restriction with or without paricalcitol in type 2 diabetes and losartan-resistant macroalbuminuria (PROCEED): a randomised, double-blind, placebo-controlled, crossover trial. Lancet Diabetes Endocrinol. 2018 Jan;6(1):27-40. doi: 10.1016/S2213-8587(17)30359-5. Epub 2017 Nov 2. PMID 29104158